CLINICAL TRIAL: NCT01656915
Title: Ex Vivo LPS Stimulation in Healthy and Compromised Subjects
Status: Completed | Type: Observational
Sponsor: TNO (Other)
Collaborators: Unilever R&D (Industry); Netherlands Metabolomic Center (NMC), The Netherlands (Unknown)
Responsible Party: Principal Investigator, W.J. Pasman, Principal Investigator, PhD, TNO
Other Study IDs: CHDR1212
Record Dates: First submitted 2012-06-20; First posted 2012-08-03 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Compromised Health; Healthy
Keywords: inflammation; response; resilience; cytokines; pre-diabetes
MeSH Terms: conditions — Inflammation; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained for standard clinical chemistry, heamatology, cytokines and ex vivo LPS stimulation.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy men: Healthy male subjects with normal weight
- Compromised men: pre-diabetic overweight, male subjects

SUMMARY:
Ex vivo LPS stimulation of whole blood will be a good alternative challenge to induce an inflammatory response and examine differences in the inflammatory response between healthy and compromised subjects.

The purpose of the current study is to examine the inflammatory response in a younger population (35-45 yrs old) to see whether in this population also differences in the ex vivo LPS induced cytokine response exists between healthy and compromised subjects, as is seen in elderly subjects. Overweight subjects showing a state of disturbed blood glucose control will be included as subjects with compromised health and compared to healthy lean subjects with the same age (shifting from healthy towards unhealthy, not diseased).

Hypothesis Ex vivo LPS stimulation of whole blood will induce a measurable inflammatory cytokine response in a healthy population that is different from a response of the compromised population. The investigators will include subjects aged 35-45 years that differ in health characteristics, especially blood HbA1c, fat% and waist circumference.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the health and lifestyle questionnaire, physical examination and results of the pre-study laboratory tests;
2. Males aged between 35-45 years;
3. Waist circumference: healthy < 94 cm, compromised ≥ 102 cm.
4. Body composition (InBody 720): body fat % healthy men < 8-19% %; for compromised men > 25%;
5. HbA1c levels for healthy subjects < 5.5 % or fasting glucose > 3.4 or < 5.6 mmol/L; for compromised HbA1c >=6 and< 6.5% or fasting glucose between 6.1-6.9 mmol/L;
6. Regular Dutch eating habits as assessed (three main meals, including bread) by health and lifestyle questionnaires.

Exclusion Criteria:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study;
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances;
3. Having a history of medical or surgical events that may significantly affect the study outcome, including any psychiatric history, and metabolic or endocrine disease, or any gastro-intestinal disorder or inflammatory diseases or allergy;
4. Use of any medication within 14 days before day 01; use of paracetamol within 7 days before day 01;
5. Currently smoking or stopped smoking less than 6 months ago;
6. Alcohol consumption >= 21 units per week;
7. Performing more than 5 hour sports activity per week;
8. Use of dietary supplements that could affect the inflammatory response (eg fish oil, polyphenols, vitamins);
9. Not having a general practitioner;
10. Not willing to accept information transfer which concerns participation in the study, or information regarding health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner;
11. Not willing to give permission to have the general practitioner to be notified upon participation in this study.

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In total, 36 male subjects will participate in the study. The study will be conducted in two different subject groups (one healthy and one compromised group), each consisting of 18 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Cytokines | baseline, 4h and 24h incubation with ex vivo LPS
  The levels of interleukines present in healthy and compromised subjects will be determined in a baseline sample.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Peeters, PhD, Principal Investigator — CHDR Leiden
Locations (1):
- CHDR, Leiden, South Holland, Netherlands

REFERENCES:
- [Background] Wijsman CA, Maier AB, de Craen AJ, van den Biggelaar AH, Westendorp RG. An unopposed proinflammatory response is beneficial for survival in the oldest old. Results of the Leiden 85-plus Study. J Gerontol A Biol Sci Med Sci. 2011 Apr;66(4):393-9. doi: 10.1093/gerona/glq212. Epub 2010 Dec 22. PMID 21177757